CLINICAL TRIAL: NCT02748317
Title: The Impact of Self-Management With Probiotics on Urinary Symptoms and the Urine Microbiome in Individuals With Spinal Cord Injury (SCI) and Spina Bifida (SB)"
Brief Title: Impact of Probiotics on Urinary Symptoms in Spinal Cord Injury SCI and SB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Georgetown University (Other); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-211
Record Dates: First submitted 2016-01-29; First posted 2016-04-22 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Spina Bifida; Spinal Cord Injury; Lower Urinary Tract Symptoms; Probiotics; Intermittent Catheterization
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Spinal Dysraphism; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adults with Spinal Cord Injury (Experimental): Lactobacillus rhamnosus GG
  Interventions: Drug: Lactobacillus rhamnosus GG

INTERVENTIONS:
Drug: Lactobacillus rhamnosus GG — For the intravesicular Lactobacillus instillation, participants will be instructed to mix the contents of 1 Lactobacillus capsule into 45 cc sterile 0.9% saline.5,6 After mixing, participants will draw up the 45 cc of the liquid Lactobacillus mixture into a 60cc catheter tip syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Participants will receive 10 Lactobacillus GG tabs at the beginning of treatment phase. At the end of each month, the coordinator or RA will ask how many remaining tablets the participant has, and if needed dispense the next supply of 10 tablets Participants will be instructed to complete the USQ-NB weekly.
  Other Names: Culturelle

SUMMARY:
As a collaborative effort between MedStar National Rehabilitation Hospital (NRH)/MedStar Health Research Institute (MHRI), Children's National Medical Center (CNMC) Department of Urology, Children's Research Institute (CRI) Center for Genetic Medicine Research, and Georgetown University Medical Center, the overall objective of this study is to develop, validate, and assess a patient-initiated, probiotics-based, self management protocol that is initiated at the time of urinary symptoms. The self-management protocol will allow patients to manage urinary symptoms and avoid potentially unnecessary antibiotic use, and provide a readily-available means of maintaining health, function, and independence throughout the lifespan.

DETAILED DESCRIPTION:
Lower urinary symptoms are a common issue for individuals with neurogenic bladder, commonly occurring in the Spina bifida and Spinal Cord Injury population. In this study, probiotics will be introduced into the bladder to prevent UTIs. Introduction of probiotics will be determined by a validated symptom questionnaire (USQ-NB) and protocol (SMP-PRO).

This study will estimate the strength of the associations between successful implementation of the probiotic self-management program (USQ-NB and SMP-PRO) and urinary symptoms, bladder inflammation, and the urine microbiome. Investigators will conduct an 18-month study in which each participant will serve as his/her own control through 3 phases of study: 6-months usual care (baseline), 6-months probiotic intervention, and 6-months follow-up.

Participants will complete the Urinary Symptom Questionnaire weekly. After 6 months of baseline data collection, participants will receive the Lactobacillus (Culturelle GG, 20 billion live organisms for adults and 10 billion live organisms for children <18 years of age), will be instructed on preparation and intravesicular instillation of the Lactobacillus, and will have a tutorial with a fellow consumer on use of the patient-initiated protocol. The protocol and Lactobacillus bladder instillation instructions (including a step-by-step video) will be available on the study website for 24/7 access and written instructions will be provided at the time of instruction.

For the intravesicular Lactobacillus instillation, participants will be instructed to mix the contents into sterile saline. After mixing, participants will draw up the liquid Lactobacillus mixture into a 60cc catheter tip syringe and instill via the intermittent catheter after fully emptying the bladder. Participants will be instructed not to catheterize for at least 4 hours after the bladder instillation. Participants will receive 10 Culturelle GG at the beginning of the treatment phase. At the end of each month, the coordinator or RA will ask how many remaining tablets the participant has, and if needed dispense the next supply of 10 tablets. Participants will be instructed to complete the USQ-NB weekly.

If/when urinary symptoms occur, subjects will be instructed to follow the protocol to determine whether to initiate intravesicular Lactobacillus instillation or be evaluated by a physician. The self-management protocol will also direct them to discontinue Lactobacillus instillation or be evaluated by a physician if symptoms remit, persist (after 2 instillations), or worsen. The maximum number of instillations is 2 over 28 hours. If participants are directed by the self-management protocol to seek medical attention or s/he feels the need for medical evaluation, s/he will be advised to obtain care as they typically would by their health care provider. Participants will be supplied with letters to be brought to their health care provider notifying them of the study and requesting sharing of urinalysis and urine culture results with the research team. A verified UTI will include those that resulted in antibiotic treatment by a health care professional. An additional urine sample for metagenomics will either be left with the health care provider for pick up by the research team, brought to the research site, or obtained by the RA at a mutually convenient site.

After completion of the 6-month patient-initiated, self-management protocol intervention period, participants will monitor symptoms weekly using the USQ-NB for the final 6-month phase of the 18-month study.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. SCI, SB or MS at least 1-year duration
3. Neuropathic bladder, as determined by the attending physician
4. Utilizing intermittent catheterization for bladder management
5. A history of 2 or more UTIs in the past year
6. Community dwelling.

Exclusion Criteria:

1. Known genitourinary pathology beyond neuropathic bladder (i.e., vesicoureteral reflux, bladder or kidney stones, etc.)
2. Use of prophylactic antibiotics
3. Instillation of intravesicular agents to reduce UTI (i.e., gentamycin)
4. Psychologic or psychiatric conditions influencing the ability to follow instructions
5. Participation in another study in which results would be confounded
6. Pregnant or breastfeeding
7. Individuals with a history of acquired or genetic immunodeficiencies; active, acute or chronic serious infections (i.g., viral hepatitides, HIV/AIDs)
8. Individuals with cancer/autoimmune disorders
9. Serious allergy to any component or excipients in the live bacterial combination product
10. No change in neurologic status in the previous 2 weeks
11. Taken antibiotic for any reason in the previous 2 weeks
12. Any patient with history of sensitivity or allergy to ampicillin or tetracycline
13. Current urinary tract infection or urinary tract infection within the previous 2 weeks (as defined by Infectious Diseases Society of America CAUTI Guidelines, 2010).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne L Groah, MD, MSPH, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited nationwide between Jan 20, 2016, and May 31, 2017
Groups:
- Adults With Spinal Cord Injury, Spina Bifida or MS: Lactobacillus instillation: During intervention phase participants were instructed to instill a Lactobacillus solution via their intermittent catheter when they experienced cloudier or more bad- smelling, stronger, fouler or more pungent than their normal urine. These symptoms had to be experienced in the absence of fever, shaking chills, feeling unclear, foggy or confused, overall sense of discomfort, feeling more tired than usual, side pain in the lower back, tenderness to touch in the side of the low back, blood in urine, abdominal pain below, belly button, increase in muscle tightness or tone, autonomic dysreflexia, sense of unease.
Period: Overall Study
Arm/Group | Adults With Spinal Cord Injury, Spina Bifida or MS
Started | 96
Completed | 73
Not Completed | 23
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 8
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Adults With Spinal Cord Injury, Spina Bifida or MS: Lactobacillus instillation During intervention phase participants were instructed to instill a Lactobacillus solution via their intermittent catheter when they experienced cloudier or more bad- smelling, stronger, fouler or more pungent than their normal urine. These symptoms had to be experienced in the absence of fever, shaking chills, feeling unclear, foggy or confused, overall sense of discomfort, feeling more tired than usual, side pain in the lower back, tenderness to touch in the side of the low back, blood in urine, abdominal pain below, belly button, increase in muscle tightness or tone, autonomic dysreflexia, sense of unease.
Arm/Group | Adults With Spinal Cord Injury, Spina Bifida or MS
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 89
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 43.7 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 18
  White | 70
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Lactobacillus Safety
Description: Total Adverse Events (AE + Serious AE) per participant .
Time Frame: months 1-18 of study
Population: All adult study participants
Measure: Mean (Standard Deviation); unit: Adverse Events
Arm/Group | Adults With Spinal Cord Injury, Spina Bifida or MS
Number analyzed (Participants) | 96
Adverse Events | .594 (1.09)
Statistical Analysis 1: Comparison: Adults With Spinal Cord Injury, Spina Bifida or MS; Test type: Other — 1 group t-test no comparison group; p = 0.219, t-test, 2 sided — P-value is not adjusted

2. Secondary Outcome: Lactobacillus Tolerability
Description: This is a one-item satisfaction rating. "While thinking only about the preceding 6-month time period: "can you estimate, using a scale from 0 to 100%, whether or not you would seek out this intervention and pay for it yourself if insurance did not pay for it?" Participants indicated their answer by moving a "slider" with three anchors: 0%=Would absolutely never do this; 50%=Might do this; 100%= Would absolutely do this. If a participant is less satisfied, their rating will be lower, and if they are more satisfied, the rating would be higher, but the item did not have options for "better" or "worse". This is not a published scale, we included this item in our general data collection.
  Ratings averaged over final 12 months of study (Satisfaction question was answered by study participants at 3 time points; 6 months, 12 months and 18 months)
Time Frame: Months 7-18
Population: 50 adult participants instilled Lactobacillus at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adults With Spinal Cord Injury, Spina Bifida or MS
Number analyzed (Participants) | 50
units on a scale | 60.6 (27.58)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected on all participants throughout their study participation which was 18 months.
Arm/Group | Adults With Spinal Cord Injury, Spina Bifida or MS
All-Cause Mortality (participants affected / at risk) | 1/96
Serious Adverse Events (participants affected / at risk) | 32/96
Other Adverse Events (participants affected / at risk) | 11/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With Spinal Cord Injury, Spina Bifida or MS (N=96)
Believed heart attack (Cardiac disorders) | 1 (1)
Sepsis/ cardiomyopathy (Cardiac disorders) | 1 (1)
Low blood pressure (Cardiac disorders) | 1 (1)
C-diff (Gastrointestinal disorders) | 1 (1)
Infection in Abcess (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Hip Infection (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fractures (Musculoskeletal and connective tissue disorders) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Mental health issues (Psychiatric disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 9 (16)
Kidney infection (Renal and urinary disorders) | 2 (2)
Prostate infection (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pressure Ulcer/ Wound (Skin and subcutaneous tissue disorders) | 2 (2) — One wound on foot, and one rectal wound
Surgery (Surgical and medical procedures) | 4 (5) — 1 Colonoscopy 1 Bladder Augmentation 1 Spinal reconstruction 1 Hysterectomy 1 Side effects hysterectomy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With Spinal Cord Injury, Spina Bifida or MS (N=96)
Physical Discomfort (General disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 6 (7)
Discomfort Instilling Lactobacillus (Renal and urinary disorders) | 1 (1)
Low urine PH value (Renal and urinary disorders) | 1 (1)
Accident with urological supplies (Social circumstances) | 1 (1)
Removal or kidney stones (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT02748317/Prot_SAP_000.pdf